CLINICAL TRIAL: NCT03593330
Title: Transitional Care Services: A Quality and Safety Process Improvement Programme in Neurosurgery
Brief Title: Neurosurgical Transitional Care Programme
Acronym: TCP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early data showed an improvement in length of stay and patient satisfaction, but the nursing time that had been provided for free was subsequently withdrawn, and it was necessary to stop the trial before sufficient data had been collected.
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Brigham and Women's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS238850; ReDA No: 012315 (Other: Joint Research Management Office)
Record Dates: First submitted 2018-06-05; First posted 2018-07-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Surgery; Brain Tumor; Brain Tumor, Recurrent; Brain Pathology; Spinal Diseases; Spinal Stenosis; Spinal Fusion; Trigeminal Neuralgia; Hydrocephalus; Fusion of Spine; Aneurysm; SPINAL Fracture; Chiari; Net; Skull Injuries; Brain Cancer; Brain Metastases; Brain Diseases; Brain Lesion; Brain Cyst; Spinal Curvature; Spinal Instability; Spinal Cord Neoplasms
Keywords: Transitional Care; Discharge Planning; Readmission; Elective Neurosurgery; Elective Spinal Surgery; Elective Brain Surgery; Transitional Care Program; TCP
MeSH Terms: conditions — Brain Neoplasms; Spinal Diseases; Spinal Stenosis; Trigeminal Neuralgia; Hydrocephalus; Aneurysm; Spinal Fractures; Brain Diseases; Spinal Curvatures; Spinal Cord Neoplasms | interventions — Patient Discharge

STUDY DESIGN:
Intervention Model Description: Patients will be randomised into two groups: standard of care or Transitional Care Programme (TCP)
Masking Description: All eligible patients will be consented to participate in the study. If they consent, a non-clinician study team member will randomise the patient into the control or intervention arm. Thereafter, all members of the care team will be notified of the patient's allocation in order to deliver the TCP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitional Care Programme (Experimental): The primary intervention of the Transitional Care Programme (TCP) will be additional patient education, framing of expectations for the hospital course and length of stay, coordinated team preparation for discharge, a dedicated discharge appointment, and a follow up phone call.
  Interventions: Other: Transitional Care Programme
- Standard of Care (No Intervention): Patients are admitted without a pre-determined discharge date. They do not receive a dedicated discharge appointment, and will not receive a follow up phone call 48 hours after discharge.

INTERVENTIONS:
Other: Transitional Care Programme — These patients will receive a pre-admission overview of their surgery, an anticipated discharge date, and a pre-scheduled discharge appointment to set patient expectations for a shorter hospitalization. On the day of discharge, the patient and his or her caregiver will attend an extended discharge appointment with a TCP-trained nurse. Finally, patients will receive a surveillance phone call 48 hours after discharge.
  Other Names: Discharge Planning
  Arms: Transitional Care Programme

SUMMARY:
Readmissions increasingly serve as a metric of hospital performance, inviting quality improvement initiatives in both medicine and surgery. Recently, a readmission reduction program in the United States was associated with significantly shorter length of stay, earlier discharge, and reduced 30-day readmission after elective neurosurgery. These results underscore the importance of patient education and surveillance after hospital discharge, and it would be beneficial to test whether the same approach yields beneficial results in a different health system, the NHS. In this study, the investigators will replicate the Transitional Care Program (TCP) with the goal of decreasing length of stay, improving discharge efficiency, and reducing readmissions in neurosurgical patients by optimizing patient education and post-discharge surveillance.

DETAILED DESCRIPTION:
Discharge Program Process Abbreviations: AA: administrative assistant; MRN: medical record number; OT: occupational therapy; PT: physical therapy; and TCT = Transitional Care Team.

CLINIC (pre-enrolment)

* Patient has clinic visit with surgeon and is identified for surgery
* Surgeon identifies that the patient is eligible to participate in the program and consents the patient for enrolment.
* Patients will be given a written information sheet on the program, and will have the opportunity to receive the information via email as well.
* Their consent will be obtained in clinic; the use of interpreters will be used for individuals with special communication needs.

AFTER CLINIC

* Once individuals consent to be randomised into the study, their MRN will be given to the TCP nurse, who will randomise the patient into the control or intervention group using a random number generator.
* Patients randomised to the TCP will be given a pre-determined discharge date when they are called to schedule their operation. The anticipated discharge date will be determined by each surgeon's expected length of stay per procedure.
* AA provides brief intro to patient about the discharge pilot, including need for family member to be present to take patient home after appointment is complete. The surgery and discharge appointments are then booked.
* AA sends surgical letter (with anticipated length of stay and discharge appointment date/time) and discharge pilot postcard to patient via email or mail
* AA enters case and discharge information into NSU Discharge Calendar
* Transitional Care Team (TCT) checks NSU Discharge Calendar daily for scheduled cases and discharge appointments

ADMISSION (TCT)

* TCT monitors operating theatre regularly for post-op pilot patients and visits daily
* TCT updates Safety Round white boards with all discharge appointment information
* TCT sends daily dept. email, including PT/OT, with following day's discharge appointment details

ADMISSION (INPATIENT/OUTPATIENT TEAMS)

* Patient is deemed appropriate for impending discharge by neurosurgery team
* TCT updates Safety Rounds white board and discusses discharge checklist with care team.
* Inpatient team completes discharge summary
* Inpatient team completes take-away medication list by 4pm one day prior to discharge appointment
* Inpatient team rationalises the need for further blood tests (as part of standard medical treatment, not for study purposes).
* Inpatient team confirms PT/OT is complete
* Inpatient team completes discharge checklist and puts in letter tray in TCP Nurse office for collection

POST-DISCHARGE APPOINTMENT

* Staff nurse or ward sister discharges patient
* TCT pulls discharge medications from pharmacy for appointments
* Healthcare assistant or staff nurse transports patient to discharge appointment
* Discharge appointment checklist completed by TCT for appointment
* Volunteer transports patient to hospital exit or Discharge Lounge

AFTER POST-DISCHARGE APPOINTMENT

* TCT/volunteer scans signed discharge appointment checklist into medical record
* TCT/volunteer records data in the spreadsheet
* TCT/volunteer shreds checklists
* TCT communicates any outstanding issues to primary teams
* Patient is asked to complete a patient satisfaction survey which will be sent via post and email. A second request will be sent at one week and two weeks post discharge.

FOLLOW-UP PHONE CALLS

* After completion of post-discharge appointments, TCT makes follow-up phone calls
* Call template is completed
* Call template is scanned into medical record
* All outstanding issues will be signed out to the primary teams by the TCT

Outcome measures will be collected through:

Intake forms Longitudinal data collection from hospital medical records and patient satisfaction surveys.

Data collected will be 30-day unplanned hospital re-admissions (to the same institution as the index operation) and length of hospital stay, the latter of which will be evaluated continuously by the number of hours of the initial hospitalisation. Time of discharge (with an early discharge defined as before 12:00 PM) will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for the TCP if scheduled for elective neurological surgery (including spinal surgery performed by an orthopedic surgeon) and were expected to have a discharge disposition to home.

Exclusion Criteria:

* Patients with an anticipated discharge to a facility other than home
* Patients with an anticipated discharge to home who are then discharged to a facility other than home will be excluded from the statistical analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | From time of hospital admission until the time of first hospital discharge or time of death from any cause, whichever came first. Assessed up to 4 months post-admission.
  Time from admission until discharge (reported in hours)

SECONDARY OUTCOMES:
Hospital Readmission | From the time of hospital discharge from the original admission until 30 days after hospital discharge
  Unplanned Readmission
Discharge before 12:00pm | This is assessed on the date of discharge from time 00:00 to time 23:59. The actual time of discharge or time of death from any cause, whichever came first, will be noted. Assessed up to 4 months post-admission.
  Early morning discharge (between 00:00 and 11:59)
Cost | The cost of the hospital admission will be calculated for the time frame from the initial hospital admission until 30 days after hospital discharge, or time of death from any cause.
  Total cost of hospital admission, transitional care programme, and readmission
Patient Satisfaction scores based on a single survey provided to the patient at the time of discharge. | From the time of hospital discharge from the original admission up until 2 weeks after discharge
  5-point Likert-scale scores will be analyzed from a single patient satisfaction survey that is provided to the patient at the time of discharge. This survey was reported previously by Robertson et al. (Journal of Neurosurgery, 2017). The patient will have 2 weeks to complete the survey. Scores will assess patient satisfaction with 1 being the least satisfied and 5 being the most satisfied. Scores will be averaged for analysis and reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Edward McKintosh, FRCS(SN) PhD, Principal Investigator — Barts Health
Locations (1):
- Bart's Health NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Robertson FC, Logsdon JL, Dasenbrock HH, Yan SC, Raftery SM, Smith TR, Gormley WB. Transitional care services: a quality and safety process improvement program in neurosurgery. J Neurosurg. 2018 May;128(5):1570-1577. doi: 10.3171/2017.2.JNS161770. Epub 2017 Jul 14. PMID 28707992
- [Background] Jones CE, Hollis RH, Wahl TS, Oriel BS, Itani KM, Morris MS, Hawn MT. Transitional care interventions and hospital readmissions in surgical populations: a systematic review. Am J Surg. 2016 Aug;212(2):327-35. doi: 10.1016/j.amjsurg.2016.04.004. Epub 2016 Jun 1. PMID 27353404
- [Background] Verhaegh KJ, MacNeil-Vroomen JL, Eslami S, Geerlings SE, de Rooij SE, Buurman BM. Transitional care interventions prevent hospital readmissions for adults with chronic illnesses. Health Aff (Millwood). 2014 Sep;33(9):1531-9. doi: 10.1377/hlthaff.2014.0160. PMID 25201657